CLINICAL TRIAL: NCT04148651
Title: Clinical Study of the CO2RE® Laser Device for Treatment of Vulvar Lichen Sclerosus
Brief Title: The CO2RE® System for Vulvar Lichen Sclerosus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Candela Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DHF25211
Record Dates: First submitted 2019-10-29; First posted 2019-11-01 (Actual); Results first posted 2021-01-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-02

CONDITIONS: Vulvar Lichen Sclerosus
Keywords: vulvar dystrophy; vulvar atrophy; persistent itching; leukoplakia; hyperkeratosis; sexual function
MeSH Terms: conditions — Vulvar Lichen Sclerosus; Leukoplakia; Keratoderma, Palmoplantar, Epidermolytic

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- CO2RE® Treatment (Experimental): All eligible subjects will undergo up to 5 treatments at 4±1-week intervals to the vulva with a fractional CO2 laser.
  Interventions: Device: The CO2RE® System

INTERVENTIONS:
Device: The CO2RE® System — The CO2RE® system is a fractional CO2 laser that is FDA-cleared under a 510(k) K181523 for laser incision, excision, ablation and/or vaporization and of soft tissue in gynecology (GYN) for the treatment of leukoplakia (vulvar dystrophies).

SUMMARY:
Subjects with vulvar lichen sclerosus (VLS) will undergo fractional carbon dioxide (CO2) laser treatment to the vulvar area. Subjects will be evaluated for changes in clinical signs and architectural changes associated with VLS at designated follow-ups to 1-year post treatment series.

DETAILED DESCRIPTION:
This study is a prospective, non-randomized, single-group assignment, interventional clinical trial. Female subjects with vulvar lichen sclerosus (VLS) supported by histologic findings on biopsy and/or clinical signs on physical examination and recalcitrant to mid- to high-potency steroid therapy, will undergo up to 5 monthly treatments to the vulva with a fractional CO2 laser.

Investigators will assess clinical signs and architectural changes associated with VLS. Baseline measurements will be compared to follow-up at 6 weeks, 3 months, 6 months and 12 months after the final treatment.

Subjects will self report sexual function using a validated FSFI Questionnaire at baseline and at the 3- and 6-month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand and sign informed consent for study participation;
2. Female subjects with age 18-80 years;
3. Biopsy demonstrates biopsy-proven lichen sclerosus and/or there are characteristic changes for vulvar lichen sclerosus on physical examination;
4. Treatment of LS has been recalcitrant to mid to high-potent topical corticosteroid treatment or subject refuses topical corticosteroid treatment. Recalcitrance to therapy is defined as no response to topical corticosteroids of an adequate potency (i.e. clobetasol propionate 0.05% ointment or other steroids) and a sufficient duration (12 weeks of use) or lack of symptomatic control of the disease with a maintenance therapy;
5. Topical corticosteroid treatment, if any, will be continued during the study period;
6. Exogenous hormone treatment, if any, will be continued during the study period (type and dose must stay consistent throughout the study);
7. One or more of the following symptoms: itch; pain unrelated to intercourse; pain, skin tearing or bleeding with intercourse; changes/decrease in sexual function;
8. No breaks, tears or lesions, malodorous discharge or strawberry cervix present on gynecological exam.

Exclusion Criteria:

1. Presence of clinically atypical appearing nevi in the area to be treated;
2. Unexplained vaginal bleeding;
3. Active infection, specifically: urinary tract infection, vulvar or vaginal infection (candidiasis, genital herpes/herpes simplex virus, bacterial vaginosis, trichomonas);
4. History of vulvar or any gynecological malignancy, as well as history of pelvic radiation therapy or stem cell transplant;
5. Pelvic organ prolapse > stage 2;
6. Pregnancy or planning pregnancy during the study;
7. Systemic treatment with immuno-modulatory drugs.
8. Use of vaginal dilators during study.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Konika P Schallen, MD, Study Director — Candela Corporation
Locations (4):
- United States (4):
  - Total Dermatology Care Center, Jacksonville, Florida
  - Center for Modern Aesthetic Medicine, Jacksonville, Florida
  - HERmd (formerly Somi Javaid M.D. & Associates), Cincinnati, Ohio
  - Lumina Med Spa, South Burlington, Vermont

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sheinis M, Selk A. Development of the Adult Vulvar Lichen Sclerosus Severity Scale-A Delphi Consensus Exercise for Item Generation. J Low Genit Tract Dis. 2018 Jan;22(1):66-73. doi: 10.1097/LGT.0000000000000361. PMID 29095746
- [Background] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Background] Thorstensen KA, Birenbaum DL. Recognition and management of vulvar dermatologic conditions: lichen sclerosus, lichen planus, and lichen simplex chronicus. J Midwifery Womens Health. 2012 May-Jun;57(3):260-75. doi: 10.1111/j.1542-2011.2012.00175.x. PMID 22594865
- [Background] Salvatore S, Leone Roberti Maggiore U, Athanasiou S, Origoni M, Candiani M, Calligaro A, Zerbinati N. Histological study on the effects of microablative fractional CO2 laser on atrophic vaginal tissue: an ex vivo study. Menopause. 2015 Aug;22(8):845-9. doi: 10.1097/GME.0000000000000401. PMID 25608269
- [Result] Stewart K, Javaid S, Schallen KP, Bartlett S, Carlson NA. Fractional CO2 laser treatment as adjunctive therapy to topical steroids for managing vulvar lichen sclerosus. Lasers Surg Med. 2022 Jan;54(1):138-151. doi: 10.1002/lsm.23476. Epub 2021 Sep 20. PMID 34541702

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Although 14 subjects enrolled, 1 subject was withdrawn from the study due to a protocol violation and 1 subject was found to be not eligible prior to her first treatment. Therefore, 12 subjects are included in this analysis.
Units Other Than Participants: Treated areas
Groups:
- CO2RE® Treatment: All eligible subjects underwent up to 5 treatments at 4±1-week intervals to the vulva with a fractional CO2 laser and maintained protocol regimen.
  The CO2RE® System: The CO2RE® system is a fractional CO2 laser that is FDA-cleared under a 510(k) K181523 for laser incision, excision, ablation and/or vaporization and of soft tissue in gynecology (GYN).
Period: Overall Study
Arm/Group | CO2RE® Treatment
Started | 12; 12 Treated areas
Completed | 10; 10 Treated areas (2 subjects did not complete the final follow-up due to COVID-19 pandemic)
Not Completed | 2; 2 Treated areas
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: Although 14 subjects enrolled, 1 subject was withdrawn from the study due to a protocol violation and 1 subject was found to be not eligible prior to her first treatment. Both are not included in the Results analysis.
Groups:
- CO2RE® Treatment: All eligible subjects that underwent up to 5 treatments at 4±1-week intervals to the vulva with a fractional CO2 laser and maintained the protocol regimen.
  The CO2RE® System: The CO2RE® system is a fractional CO2 laser that is FDA-cleared under a 510(k) K181523 for laser incision, excision, ablation and/or vaporization and of soft tissue in gynecology (GYN) for treatment of leukoplakia (vulvar dystrophies).
Arm/Group | CO2RE® Treatment
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.6 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 10
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12
FSFI [Mean (Standard Deviation); unit: score on a scale] — The validated Female Sexual Function Index (FSFI) was used to compare sexual function to baseline. FSFI score, a 19-item validated questionnaire assesses domains of sexual function, including desire, arousal, lubrication, orgasm, satisfaction, and pain, in addition to providing an overall score regarding sexual function. The aggregated FSFI score is a sum of weighted answers for each of the 19 items in the questionnaire with a maximum score 36.0 (high level of sexual functional) and minimum score of 2.0 (low level of sexual functional).
  score on a scale | 13.9 (10.1)

OUTCOME MEASURES:

1. Primary Outcome: Average Scores for VLS Clinical Signs Present At Baseline, 3, 6 and 12 Months After the Last Treatment as Assessed by the Investigators
Description: Each clinical sign of VLS (loss of elasticity, sclerosis, lichenification, whitening, parchment-like skin, fissures, extent of the disease, erosions, ulcerations, hyperkeratosis, excoriation, telangiectasia) was assessed separately by the investigator, using a 4-point scale (0=not present, 1=mild, 2=moderate or 3=severe) for each subject at baseline and follow-ups. For those clinical signs present at baseline (baseline score >0 on severity scale), an average severity grade was calculated at each endpoint to evaluate overall treatment outcome, as follows:
  Average severity grade = Sum of all severity grades (0, 1, 2, or 3) for each individual parameter of clinical signs present at baseline for each subject / Number of grades
  A lower average score means better outcome.
Time Frame: At Baseline, 3, 6 and 12 months after the final treatment
Population: At Baseline, 12 subjects had 96 clinical signs present (score >0). One subject missed the 12-month follow-up, one subject missed the 3- and 12-month follow-ups and one subject missed the 6-month follow-up. Hence, at 3- and 6-month follow-up visits 11 subjects were assessed (with 89 clinical signs averaged for each visit) and at the 12-month follow-up visit 10 subjects were assessed (with 79 clinical signs averaged).
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Clinical signs
Groups:
- CO2RE® Treatment: All eligible subjects that underwent up to 5 treatments at 4±1-week intervals to the vulva with a fractional CO2 laser and maintained the protocol regimen.
  The CO2RE® System: The CO2RE® system is a fractional CO2 laser that is FDA-cleared under a 510(k) K181523 for laser incision, excision, ablation and/or vaporization and of soft tissue in gynecology (GYN).
Arm/Group | CO2RE® Treatment
Number analyzed (Participants) | 12
Number analyzed (Clinical signs) | 96
score on a scale
  Average score of clinical signs at Baseline | 1.85 (0.73)
  Average score of clinical signs at 3-months follow-up visit: number analyzed (Participants) | 11
  Average score of clinical signs at 3-months follow-up visit: number analyzed (Clinical signs) | 89
  Average score of clinical signs at 3-months follow-up visit | 0.65 (0.74)
  Average score of clinical signs at 6-months follow-up visit: number analyzed (Participants) | 11
  Average score of clinical signs at 6-months follow-up visit: number analyzed (Clinical signs) | 89
  Average score of clinical signs at 6-months follow-up visit | 0.65 (0.76)
  Average score of clinical signs at 12-months follow-up visits: number analyzed (Participants) | 10
  Average score of clinical signs at 12-months follow-up visits: number analyzed (Clinical signs) | 79
  Average score of clinical signs at 12-months follow-up visits | 0.73 (0.83)

2. Primary Outcome: Average Scores for VLS Architectural Changes Present At Baseline and at 3, 6 and 12 Months After the Last Treatment as Assessed by the Investigators
Description: Each architectural change of VLS (labial fusion, clitoral hood fusion, narrowing of the introitus, anterior changes, perianal involvement, formation of posterior commissure bands) was assessed separately by the investigator, using a 4-point scale (0=not present, 1=mild, 2=moderate or 3=severe) for each subject at baseline and follow-ups. For those architectural changes present at baseline (baseline score >0 on severity scale), an average severity grade was calculated at each endpoint to evaluate overall treatment outcome, as follows:
  Average severity grade = Sum of all severity grades (0, 1, 2, or 3) for each individual parameter of architectural changes present at baseline for each subject / Number of grades
  A lower average score means better outcome.
Time Frame: Baseline, 3 , 6 and 12 months after the final treatment
Population: At Baseline, 12 patients had 55 architectural changes present (score >0). One subject missed the 12-month follow-up, one subject missed the 3- and 12-month follow-ups and one subject missed the 6-month follow-up. Hence, at the 3- and 6-month follow-ups, 11 subjects were assessed (with 51 architectural changes averaged for each visit) and at the 12-month follow-up 10 subjects were assessed (with 49 architectural changes averaged).
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Architectural Changes
Arm/Group | CO2RE® Treatment
Number analyzed (Participants) | 12
Number analyzed (Architectural Changes) | 55
score on a scale
  Average score of architectural changes at Baseline | 2.18 (0.72)
  Average score of architectural changes at 3-month follow-up: number analyzed (Participants) | 11
  Average score of architectural changes at 3-month follow-up: number analyzed (Architectural Changes) | 51
  Average score of architectural changes at 3-month follow-up | 1.10 (0.90)
  Average score of architectural changes at 6-month follow-up: number analyzed (Participants) | 11
  Average score of architectural changes at 6-month follow-up: number analyzed (Architectural Changes) | 51
  Average score of architectural changes at 6-month follow-up | 1.04 (0.87)
  Average score of architectural changes at 12-month follow-up: number analyzed (Participants) | 10
  Average score of architectural changes at 12-month follow-up: number analyzed (Architectural Changes) | 49
  Average score of architectural changes at 12-month follow-up | 1.08 (0.91)

3. Secondary Outcome: Change From Baseline in Sexual Function on the Female Sexual Function Index (FSFI) at 3 Months and 6 Months After the Final Treatment
Description: Female Sexual Function Index (FSFI) is a validated, self-reported 19-item questionnaire that assesses domains of sexual function, including desire, arousal, lubrication, orgasm, satisfaction, and pain. The aggregated FSFI score is a sum of weighted answers for each of the 19 items in the questionnaire, with a maximum total score possible of 36.0 (high level of sexual functional) and minimum score of 2.0 (low level of sexual functional). Change = (Follow-up score - Baseline score). Mean change was calculated for all scores at the 3- and 6-month follow-ups.
Time Frame: Baseline and 3 months and 6 months after the final treatment
Population: At Baseline, 12 patients completed FSFI questionnaires. At the 3-month visit, 11 subjects completed the FSFI (one subject missed the visit). At the 6-month follow-up, 12 subjects completed the FSFI (one subject missed her visit but provided her self-assessments remotely).
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CO2RE® Treatment
Number analyzed (Participants) | 12
units on a scale
  Mean Change in FSFI At the 3-Month Follow-up: number analyzed (Participants) | 11
  Mean Change in FSFI At the 3-Month Follow-up | 4.06 (2.25)
  Mean Change in FSFI At the 6-Month Follow-up | 4.53 (2.41)

4. Secondary Outcome: Subject Satisfaction At the 12-Month Follow-up
Description: Evaluate Subject satisfaction at the 12 months post-last treatment visit, using a satisfaction scale [(-2) Very dissatisfied, (-1) Dissatisfied, (0) Uncertain, (1) Satisfied, (2) Very satisfied]. The analysis quantify the percentage of Subject satisfaction (score 1 or 2) at the 12-month follow-up.
Time Frame: 12 months after the final treatment
Population: Two subjects missed the 12-month follow-up. Therefore, subject assessments were reported for 10 subjects at the 12-month follow-up.
Measure: Count of Participants; unit: Participants
Groups:
- Subjects Treated With CO2RE® Treatment: All eligible subjects who underwent laser treatments at 4±1-week intervals to the vulva with a fractional CO2 laser and maintained the protocol regimen.
Arm/Group | Subjects Treated With CO2RE® Treatment
Number analyzed (Participants) | 10
Participants | 8

5. Secondary Outcome: Treatment Associated Pain Score
Description: Subjects underwent 3-5 monthly treatments and reported discomfort associated with treatment on a 10-cm visual analogue scale (VAS) of 0 = no pain to 10 = worst possible pain, immediately after each treatment. The outcome presented here is the mean grade of discomfort/pain associated with all treatments. Lower value presents lower treatment-associated discomfort. Since patients received 3-5 monthly treatments these values were collected at each treatment over a period of 2 to 4 months for each patient.
Time Frame: Immediately after the 1st, 2nd, 3rd, 4th and 5th monthly treatments post baseline
Population: A total of 57 sessions were conducted (10 subjects had 5 treatments,1 subject had 4 treatments and 1 subject had 3 treatments)
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Number of Treatments
Arm/Group | CO2RE® Treatment
Number analyzed (Participants) | 12
Number analyzed (Number of Treatments) | 57
score on a scale | 2.6 (2.5)

ADVERSE EVENTS:
Time Frame: The period of time over which adverse event data were collected is from treatment visit until 12-month follow-up (16 month post last treatment).
Description: The number and severity of adverse events following each treatment were evaluated at each treatment visit and at the follow-up visit up to 12 months after the last treatment.
Arm/Group | Subjects Treated With CO2RE® Treatment
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

LIMITATIONS AND CAVEATS:
Small sample size of subjects enrolled and analyzed due to delayed start at one clinical site and COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/51/NCT04148651/Prot_000.pdf